CLINICAL TRIAL: NCT00745901
Title: An Open Label Study to Evaluate Cycle Control With Ortho Tri-Cyclen Lo (Norgestimate/Ethinyl Estradiol) and Yaz (Drospirenone/Ethinyl Estradiol) in Healthy Sexually Active Females
Brief Title: Study to Evaluate Cycle Control With Norgestimate/Ethinyl Estradiol and Drospirenone/Ethinyl Estradiol in Healthy Sexually Active Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015055
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2010-05-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2012-12

CONDITIONS: Contraception
Keywords: contraception; bleeding; cycle control
MeSH Terms: conditions — Hemorrhage | interventions — norgestimate; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

INTERVENTIONS:
Drug: Norgestimate/ethinyl estradiol; Drospirenone/ethinyl estradiol

SUMMARY:
The purpose of this study in healthy sexually active females is to evaluate the cycle control with norgestimate/ethinyl estradiol versus drospirenone/ethinyl estradiol.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled, multicenter study in healthy sexually active females to evaluate cycle control with norgestimate/ethinyl estradiol versus drospireneone/ethinyl estradiol. The Open-Label Treatment Phase will last for three 28-day cycles. Approximately 300 patients will be randomized in a 1:1 fashion according to a predetermined randomization schedule. Patients will be seen for a baseline visit (Visit 1) up to 35 days prior to dosing to obtain informed consent, have a physical examination including a breast exam, height and weight, vital signs, a Chlamydia test and a urine pregnancy test performed, and to give their medical history. Patients will be instructed to report bleeding data using an interactive voice response system (IVRS) based diary on a daily basis. Patients will be instructed to continue taking 1 pill each day for 3 cycles, record this information daily in the IVRS and to contact the study site if they have any questions or adverse events they would like to discuss. The final study visit (Visit 2) will occur on Day 8 after completing 3 cycles of study medication. Patients will be weighed, have vital signs performed, report any adverse events and or changes in concomitant medications, and complete the satisfaction questionnaire at the final visit. Safety will be assessed by physical examinations, adverse events, body weight and vital signs. Patients randomized to drospireneone/ethinyl estradiol and taking any medication that could increase serum potassium levels (as outlined in the Package Insert) will also have their potassium level checked during their first cycle of treatment (Days 15 to 28 of treatment). Three 28-day cycles of either norgestimate/ethinyl estradiol or drospirenone/ethinyl estradiol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females who want oral contraception
* No cervical or vaginal abnormalities on gynecological examination
* Negative Chlamydia test
* Pap smear without evidence of moderate or severe dysplasia or any malignancy within the preceding 12 months
* Negative urine pregnancy test conducted during Visit 1
* One normal menstrual period in 35 days prior to Visit 1
* Regular menstrual cycles (every 26-35 days)
* Last term pregnancy at least 42 days prior to Visit 1, and have had at least one normal menstrual period (typical in duration and amount of flow for the subject) since her last pregnancy
* Post-menarcheal and pre-menopausal
* At least one normal menstrual period (typical in duration and amount of flow for the subject) since having undergone uterines urgery or removal of an IUD, Norplant, DepoProvera or other hormonal injectables or implants.

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to steroid hormonal therapy
* Previously discontinued ORTHO TRI-CYCLEN LO or YAZ due to breakthrough bleeding
* Pregnant or lactating
* Body mass index (BMI) of >40kg/m2
* Clinical evidence of carcinoma or other malignancy (history of basal cell carcinoma of the skin is not exclusionary)
* History of alcohol or drug abuse in the investigator's judgment based on history and physical examination (within 12 months prior to Visit 1)
* Significant depression or psychiatric disease in the investigator's judgment based on history and physical examination which would result in an unreliable patient
* Patient deemed by the investigator to have questionable reliability in her ability to comply with the protocol and provide accurate information
* Have any medical condition or planned surgical procedure which, in the opinion of the investigator, may be exacerbated by treatment with study medication or a patient receiving any concurrent therapy that could be affected by treatment with study medication
* Disallowed therapies: currently taking therapeutic anticoagulants (e.g,. Coumadin, Heparin) or have a bleeding disorder (e.g. von Willebrand's Disease), DepoProvera or other hormonal injectables in the six months before Visit 1, currently have Norplant or other hormonal implants in place, or have had removal of Norplant within 60 days prior to Visit 1, used a steroid-containing IUD within 3 months prior to Visit 1
* Or current use of an IUD
* Consistently elevated blood pressure defined as sitting systolic BP>140 mmHg or diastolic BP>90 mmHg
* Have an untreated thyroid disorder in the investigator's judgment based on history and physical examination
* unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Patients who in the opinion of the investigator should not be enrolled in the study based on the product labeling for ORTHO TRI-CYCLEN LO and YAZ including potential drug-drug interactions
* Have received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Result] Kaunitz AM, Burkman RT, Fisher AC, LaGuardia KD. Cycle control with a 21-day compared with a 24-day oral contraceptive pill: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1205-1212. doi: 10.1097/AOG.0b013e3181beab47. PMID 19935020
- See also: An Open-Label Study to Evaluate Cycle Control with ORTHO TRI-CYCLEN LO (norgestimate/ethinyl estradiol) and YAZ (drospirenone/ethinyl estradiol) in Healthy, Sexually Active Females — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=37&filename=CR015055_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- NGM/25mcg EE: NGM=norgestimate; EE=ethinyl estradiol. Days 1-7: 180 mcg NGM/25 mcg EE; Days 8-14: 215 mcg NGM/25 mcg EE; Days 15-21: 250 mcg NGM/25 mcg EE; Days 22-28: inert ingredients
- DRSP/20mcg EE: DRSP=drospirenone; EE=ethinyl estradiol. Days 1-24: 3 mg DRSP/20 mcg EE; Days 25-28: inert ingredients
Period: Overall Study
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Started | 178 (Number of Patients Randomized) | 177 (Number of Patients Randomized)
Completed | 154 | 156
Not Completed | 24 | 21
Not completed — Adverse Event | 3 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 7 | 4
Not completed — Pregnancy | 2 | 4
Not completed — Lack of compliance | 2 | 2
Not completed — Patient's next menses did not start with | 1 | 0
Not completed — Results of Pap smear at Vis 1 malignant | 0 | 2
Not completed — Chlamydia test at Visit 1 was positive | 1 | 1
Not completed — Patient didn't take any study medication | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE | Total
Number analyzed (Participants) | 178 | 177 | 355
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  >= 18 and < 65 years | 178 | 177 | 355
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.70) | 27.2 (6.52) | 27.2 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 177 | 355
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Days of Unscheduled Blood Loss - Cycle 1
Description: cycle control between treatment groups, cycle 1. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Unscheduled bleeding is any bleeding during active pills except days 1-4 of cycle 2 or 3 if contiguous with withdrawal bleeding and days 1-7 of the first cycle.
Time Frame: Cycle 1 (Day 8 to 21 for NGM/25mcg EE and day 8 to 24 for DRSP/20mcg EE)
Population: Efficacy Analysis Population: all randomized patients who took study drug and for whom there was post-baseline blood loss data after Day 7.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 1.9 (3.14) | 2.0 (3.53)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.9698, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Patient Satisfaction - Overall
Description: patient satisfaction based on 5 questions during three 28-day cycles - Question 1 (Overall Satisfaction). On a scale of 1 to 5 where 1=Very satisfied and 5=Very dissatisfied.
Time Frame: Cycle 1 to Cycle 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Participants
  Number of responses | 159 | 162
  1. Very Satisfied | 99 | 115
  2. Somewhat satisfied | 35 | 32
  3. Neither satisfied or dissatisfied | 12 | 6
  4. Dissatisfied | 11 | 8
  5. Very dissatisfied | 2 | 1
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0715, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Days of Unscheduled Blood Loss - Cycle 2
Description: cycle control between treatment groups, cycle 2. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Unscheduled bleeding is any bleeding during active pills except days 1-4 of cycle 2 or 3 if contiguous with withdrawal bleeding and days 1-7 of the first cycle.
Time Frame: Cycle 2 (Day 29 to 49 for NGM/25mcg EE and day 29 to 52 for DRSP/20mcg EE)
Population: Efficacy Analysis Population: all randomized patients who took study drug and for whom there was post-baseline blood loss data after Day 7. Include patients with at least one day evaluable in cycle 2.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 160 | 165
Days | 1.3 (2.49) | 1.9 (2.86)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0050, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Number of Days of Unscheduled Blood Loss - Cycle 3
Description: Number of Days of Unscheduled Blood Loss - Cycle 3. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Unscheduled bleeding is any bleeding during active pills except days 1-4 of cycle 2 or 3 if contiguous with withdrawal bleeding and days 1-7 of the first cycle.
Time Frame: Cycle 3 (Day 57 to 77 for NGM/25mcg EE and day 57 to 80 for DRSP/20mcg EE)
Population: Efficacy Analysis Population: all randomized patients who took study drug and for whom there was post-baseline blood loss data after Day 7. Include patients with at least one day evaluable in cycle 3.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 157 | 159
Days | 1.4 (2.33) | 2.4 (2.86)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0006, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Overall Number of Days of Unscheduled Blood Loss
Description: cycle control between treatment groups, for three 28-day cycles. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Unscheduled bleeding is any bleeding during active pills except days 1-4 of cycle 2 or 3 if contiguous with withdrawal bleeding and days 1-7 of the first cycle.
Time Frame: Cycle 1 to Cycle 3 (Day 8 to Day 80)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 4.6 (5.33) | 6.1 (6.07)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0031, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Number of Participants With the Indicated Number of Unscheduled Blood Loss Episodes
Description: Unscheduled blood loss episodes are bounded on both sides by at least 1 non- bleeding day.
Time Frame: Cycle 1 to Cycle 3 (Day 8 to Day 80)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Participants
  0 Episode | 55 | 29
  1 Episode | 46 | 41
  2 Episodes | 23 | 50
  3 Episodes | 21 | 22
  4 Episodes | 13 | 11
  5 Episodes | 7 | 8
  6 Episodes | 0 | 2
  8 Episodes | 0 | 3
  9 Episodes | 0 | 1
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0013, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Number of Days of Scheduled Blood Loss - Cycle 1
Description: cycle control between treatment groups, cycle 1. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Scheduled bleeding was defined as any bleeding that occurred while not taking active hormones, regardless of the duration of regimen.
Time Frame: Cycle 1 (Day 22 to 32 for NGM/25mcg EE and day 25 to 32 for DRSP/20mcg EE)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 4.3 (2.09) | 3.2 (2.35)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Number of Days of Scheduled Blood Loss - Cycle 2
Description: cycle control between treatment groups, cycle 2. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Scheduled bleeding was defined as any bleeding that occurred while not taking active hormones, regardless of the duration of regimen.
Time Frame: Cycle 2 (Day 50 to 60 for NGM/25mcg EE and day 53 to 60 for DRSP/20mcg EE)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 160 | 165
Days | 4.0 (2.15) | 2.8 (2.40)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Number of Days of Scheduled Blood Loss - Cycle 3
Description: cycle control between treatment groups, cycle 3. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Scheduled bleeding was defined as any bleeding that occurred while not taking active hormones, regardless of the duration of regimen.
Time Frame: Cycle 3 (Day 78 to 84 for NGM/25mcg EE and day 81 to 84 for DRSP/20mcg EE)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 157 | 159
Days | 3.1 (2.09) | 1.2 (1.30)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Overall Number of Days of Scheduled Blood Loss
Description: summary of the overall number of days of scheduled blood loss. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity. Scheduled bleeding was defined as any bleeding that occurred while not taking active hormones, regardless of the duration of regimen.
Time Frame: Cycle 1 to Cycle 3 (Day 8 to Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 11.2 (5.40) | 7.0 (4.80)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Number of Days of Total Blood Loss - Cycle 1
Description: cycle control between treatment groups, cycle 1. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity.
Time Frame: Cycle 1 (Day 8 to Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 6.2 (3.88) | 5.2 (4.45)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0033, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Number of Days of Total Blood Loss - Cycle 2
Description: cycle control between treatment groups, cycle 2. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity.
Time Frame: Cycle 2 (day 29 to Day 56)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 160 | 165
Days | 5.3 (2.66) | 4.6 (3.25)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.0060, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Number of Days of Total Blood Loss - Cycle 3
Description: cycle control between treatment groups, cycle 3. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity.
Time Frame: Cycle 3 (Day 57 to Day 84)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 157 | 159
Days | 4.6 (2.64) | 3.6 (3.10)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Overall Number of Days of Total Blood Loss
Description: cycle control between treatment groups, overall. Cycle control includes number of days of blood loss, incidence of blood loss, number of blood loss episodes, and blood loss flow intensity.
Time Frame: Cycle 1 to 3 (Day 8 to Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Days | 15.8 (6.58) | 13.2 (6.90)
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Number of Participants With Unscheduled Bleeding Cycle 1
Description: Unscheduled bleeding is any bleeding during active pills except days 1-4 of cycle 2 or 3 if contiguous with withdrawal bleeding and days 1-7 of the first cycle.
Time Frame: Cycle 1 (Day 8 to 21 for NGM/25mcg EE and day 8 to 24 for DRSP/20mcg EE)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Participants | 72 | 74
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.912, Fisher Exact

16. Primary Outcome: Number of Participants With Unscheduled Bleeding Cycle 2
Description: as for outcome 15
Time Frame: Cycle 2 (Day 29 to 49 for NGM/25mcg EE and day 29 to 52 for DRSP/20mcg EE)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 160 | 165
Participants | 57 | 87
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.003, Fisher Exact

17. Primary Outcome: Number of Participants With Unscheduled Bleeding Cycle 3
Description: as for outcome 15
Time Frame: Cycle 3 (Day 57 to 77 for NGM/25mcg EE and day 57 to 80 for DRSP/20mcg EE)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 157 | 159
Participants | 65 | 94
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.002, Fisher Exact

18. Primary Outcome: Number of Participants With Breakthrough Bleeding/Spotting Cycle 1
Description: Breakthrough bleeding/spotting is any bleeding or spotting during active pills excluding days contiguous with withdrawal bleeding or continual withdrawal bleeding.
Time Frame: Cycle 1 (Day 8 to 21 for NGM/25mcg EE and day 8 to 24 for DRSP/20mcg EE)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 165 | 167
Participants | 53 | 56
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.816, Fisher Exact

19. Primary Outcome: Number of Participants With Breakthrough Bleeding/Spotting Cycle 2
Description: as for outcome 18
Time Frame: Cycle 2 (Day 29 to 49 for NGM/25mcg EE and day 29 to 52 for DRSP/20mcg EE)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 160 | 165
Participants | 39 | 62
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.012, Fisher Exact

20. Primary Outcome: Number of Participants With Breakthrough Bleeding/Spotting Cycle 3
Description: as for outcome 15
Time Frame: Cycle 3 (Day 57 to 77 for NGM/25mcg EE and day 57 to 80 for DRSP/20mcg EE)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Number analyzed (Participants) | 157 | 159
Participants | 47 | 74
Statistical Analysis 1: Comparison: NGM/25mcg EE vs DRSP/20mcg EE; Test type: Superiority or Other; p = 0.003, Fisher Exact

ADVERSE EVENTS:
Time Frame: 35 days prior to the first day study drug was taken to study day 91 (or 7 days after last day of study drug)
Description: Total participants at risk is based on safety population, which is defined as participants who took at least one dose of study drug. Based on this definition, the total participants at risk are 167 for each of the two treatment groups.
Arm/Group | NGM/25mcg EE | DRSP/20mcg EE
Serious Adverse Events (participants affected / at risk) | 2/167 | 1/167
Other Adverse Events (participants affected / at risk) | 34/167 | 34/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NGM/25mcg EE (N=167) | DRSP/20mcg EE (N=167)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Pelvic hemorrhage (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NGM/25mcg EE (N=167) | DRSP/20mcg EE (N=167)
Acne (Skin and subcutaneous tissue disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Breast tenderness (Reproductive system and breast disorders) | 2 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1
Irritability (General disorders) | 1 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Liposuction (Surgical and medical procedures) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Mood swings (Psychiatric disorders) | 3 | 5
Migraine (Nervous system disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 3 | 0
Palpitations (Cardiac disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 1
Pelvic hemorrhage (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tension headache (Nervous system disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal cyst (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Vulval abscess (Infections and infestations) | 1 | 0
Weight increased (Investigations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less